CLINICAL TRIAL: NCT02276989
Title: Evaluation of a Compliance Marker A Supplement to: U01DA029580-02 Opioid-Induced Hyperalgesia In Prescription Opioid Abusers: Effects of Pregabalin
Brief Title: Evaluation of a Compliance Marker in Prescription Opioid Abusers With Chronic Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Peggy Compton, Professor and Associate Dean, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-0751
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Compliance; Chronic Pain
Keywords: Chronic Pain; Compliance Marker; Narcotic Abuse; Opioid related disorders; Opiate substitution treatment; Buprenorphrine; Suboxone; Lyrica; Pregabalin; Acetazolamide; Quinine; Compliance
MeSH Terms: conditions — Patient Compliance; Chronic Pain; Narcotic-Related Disorders; Opioid-Related Disorders | interventions — Acetazolamide; Quinine; Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Compliance Intervention (Experimental): Subjects will receive acetazolamide, quinine and riboflavin as experimental compliance markers and will serve as their own controls.
  Interventions: Drug: acetazolamide; Drug: Quinine; Drug: Riboflavin

INTERVENTIONS:
Drug: acetazolamide — On evening of Day 0, subjects will arrive at the session previously stabilized on buprenorphine and pregabalin. Pregabalin titration = 6 days prior to Day 0, during which time they will receive 100mg/day x 2 days, 200mg/day x2 days, and 300mg/day x 2 days, with the subjects receiving the full dose of 400mg/day beginning Day 0.
  On Day 1, pregabalin PK measures will be collected.
  On the mornings (8am) of Days 1 - 5, PGB compounded with the first tracer, ACZ will be administered.
  On Day 5, subjects will again undergo PK testing on PGB + ACZ tracer.
  On Day 6, subjects will be administered PGB and ACZ compounded with RIBO, and PK measures again collected.
  On the mornings of Days 7-8 subjects will receive their PGB dose only.
  Other Names: ACZ
Drug: Quinine — On the morning of Days 8-11, subjects will be administered the same dose of PGB, now compounded with the QUIN.
  On Day 11, PK testing of QUIN and PGB will be repeated.
  On Day 12, subjects will be administered PGB and QUIN compounded with RIBO, and PK measures again collected.
  On Day 13 patients will be discharged with take-home doses of PGB that will taper to zero over the period of one week.
  Other Names: QUIN
Drug: Riboflavin — All subjects will receive riboflavin on the following days of the study:
  On Day 6, subjects will be administered PGB and ACZ compounded with RIBO, and PK measures again collected.
  On Day 12, subjects will be administered PGB and QUIN compounded with RIBO, and PK measures again collected.
  Other Names: Vitamin B2

SUMMARY:
In a small, well-characterized sample of prescription opioid abusers (POAs) with chronic pain and on buprenorphine therapy, this study will investigate the utility and feasibility of two novel tracer compounds, and in combination with a standard marker (riboflavin), to monitor adherence to study drug prescription in the parent clinical trial.

DETAILED DESCRIPTION:
In a small, well-characterized sample of prescription opioid abusers (POAs) with chronic pain and on buprenorphine therapy, this supplement study will investigate the utility and feasibility of two novel tracer compounds, and in combination with a standard marker (riboflavin), to monitor adherence to study drug prescription in the parent clinical trial (NCT01821430).

1. We will examine the ability of two benign (in the doses used) medications, quinine (80mg) and acetazolamide (15mg) to serve as valid and reliable markers of medication use. The relative utility of each will be described for use with the study medication (PGB 400mg/day), a drug dependent on primarily renal excretion. In that both PGB and acetazolamide are eliminated unchanged in the urine, we will examine if the latter can be used without altering the elimination rate of the former, or whether a maker with both hepatic and renal modes of elimination (quinine) would serve as a better indicator of adherence in the trial.
2. Being a standard in clinical trials, the medication adherence marker riboflavin is used in the parent study (NCT01821430), as it can be readily detected in urine samples by simple visual inspection. However, riboflavin is a relatively gross indicator of medication use; it does not reside in the body for the time period typically required in outpatient trials, can be affected by dietary riboflavin and has variable absorption. Capitalizing on riboflavin's ease of detection, the second aim of this supplement will be to examine whether riboflavin when combined with one of the new candidate tracers, can provide a superior indicator of adherence, in that riboflavin can be qualitatively observed immediately, and the other tracer being quantitatively detected during subsequent urine toxicology analyses.

The cross over design of the study will allow us to address these aims in an efficient and straightforward manner. Following examination of the pharmacokinetics (PK) of PGB alone, it's PK will then be reexamined when compounded with acetazolamide, and again with both acetazolamide and riboflavin present. Next, after a short washout period, the studies PGB PK will be repeated with acetazolamide replaced by quinine. If the new tracers do not interfere with the PK of PGB, one of them will be chosen to be formulated (along with riboflavin) with PGB for use in the parent study, thereby providing both qualitative and quantitative indicators of adherence.

ELIGIBILITY:
Inclusion Criteria:

1. male and female English-speaking literate adults age 18- 50 years old,
2. have medically diagnosed chronic pain condition,
3. be on a stable dose of buprenorphine (clinic modal dose),
4. history of prescription opioid abuse,
5. adequate venous access,
6. if female, a negative pregnancy test. Individuals will not be accepted who are unstable in buprenorphine treatment as evidence by continued illicit drug use and irregular clinic attendance in the previous trial,
7. be otherwise in good physical health or in care of a physician who is wiling to take responsibility for such treatment. The same conditions apply in cases of patients with a psychiatric disorder needing ongoing treatment.

Exclusion Criteria:

1. physiologic drug dependence on benzodiazepines, barbiturates, and/or alcohol that would require medical management,
2. significant ongoing medical problems (e.g., diabetes),
3. history of head injury or seizure,
4. serious psychiatric illness outside of drug use (e.g., schizophrenia),
5. recent use of any agent that inhibits or induces cytochrome P450 3A4 or 2D6,
6. nursing or pregnant female, or a female or male who does not agree to not become pregnant or father a child during the course of, and three months following completion of the study,
7. have a cardiac conduction or blood clotting disorder,
8. blood donation within the past 30 days prior to screening,
9. clinically significant laboratory results (as judged by the investigator/sub-investigator)
10. moderate to severe COPD,
11. renal impairment, and
12. severe renal hepatic impairment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profiles for each medication/tracer (assayed from blood and urine samples) and will include parameters such as AUC, CMAX, TMax, and t1/2. | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Compton, RN, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States